CLINICAL TRIAL: NCT05914168
Title: Clinical Data Collection in Breast Tomosynthesis: COBRIS
Brief Title: Clinical Data Collection in Breast Tomosynthesis (COBRIS)
Acronym: COBRIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 179549298
Record Dates: First submitted 2022-12-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Subjects with investigational acquisition
  Interventions: Device: Breast Tomosynthesis

INTERVENTIONS:
Device: Breast Tomosynthesis — Three dimensional mammography

SUMMARY:
The purpose of the study is to assess an image acquisition application for breast tomosynthesis in a clinical environment

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo their routine mammography examination. One additional mammography view will be obtained with the investigational application and analyzed. Subject participation is expected to last no more than 30 minutes. After the mammography examination, subjects will be followed according to the hospital standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 35 years or older;
* Women referred for unilateral or bilateral 2D and 3D mammography;
* Women able and willing to comply with study procedures;
* Women able and willing to participate in this study who have signed and dated the informed consent form; and
* Women surgically sterile or postmenopausal or, the possibility of pregnancy is ruled out based on a negative urine pregnancy test

Exclusion Criteria:

* Women who have been previously included in this study; or
* Be a minor, protected adult, adult deprived of liberty by judicial or administrative decision, pregnant, parturient or a breastfeeding mother; or
* Women with BRCA 1 or BRCA 2 gene mutation

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 150 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Data Collection | 1 year
  Collect clinical breast images obtained with the investigational application.

SECONDARY OUTCOMES:
Assessment of Image Quality | 1 year
  Assess image quality through subjective and open expert evaluation of patient motion, visibility of replication artefacts and visibility of clinical findings.

CONTACTS AND LOCATIONS:
Overall Officials: Balleyguier, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No